CLINICAL TRIAL: NCT04463433
Title: Psychological Intervention for Parent-child Relationship and Couple Relationship Under COVID-19 in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Normal University (Other)
Responsible Party: Principal Investigator, Xiuyun Lin, professor, Beijing Normal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: bnulxy
Record Dates: First submitted 2020-04-12; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Parent-child Relationship and Couple Relationship Under COVID-19 in China
Keywords: COVID-19; Parent-child Relationship; Couple Relationship
MeSH Terms: conditions — COVID-19 | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent-child Relationship Intervention (Experimental): The intervention involves five 2h weekly group sessions in which exercises in mindfulness are practiced and associated ABCDE theory is taught to improve emotional regulation and parent-child communication under COVID-2019.
  Interventions: Behavioral: Cognitive and behavioral intervention.
- Couple Relationship Intervention (Experimental): The intervention involves four 2h weekly group sessions in which express feelings and wants clearly are practiced and associated Satir communication model is taught to improve couple conflict resolution and communication under COVID-2019.
  Interventions: Behavioral: Problem-solving and relationship improvement intervention.

INTERVENTIONS:
Behavioral: Cognitive and behavioral intervention. — Two hours group sessions including mindfulness and emotion regulation. The practice of mindfulness is taught to parents to become aware of their thoughts and emotion on the present moment. The behavioral intervention has parents develop an Positive Time-out for dealing with conflict and negativity, using strategies to down-regulate their own negative emotions.
  Arms: Parent-child Relationship Intervention
Behavioral: Problem-solving and relationship improvement intervention. — Two hours group sessions including problem-solving and improving marital relationship . In the problem-solving part, the knowledge and techniques of problem-solving are taught to couple. relationship improvement part which promote the couple relationship by being aware of their own and their partner's deep-seated needs and communicating in a congruent way.
  Arms: Couple Relationship Intervention

SUMMARY:
Under the COVID-19, individuals who were home Quarantine experienced new challenges on their parent-child relationship and couple relationship. The current project aimed to provide psychological interventions for both parents and couples in order to improving their relationship. The online intervention of group intervention and individual intervention are going to be conducted. The relationship between parent-child, couples and emotion regulation will be tested.

ELIGIBILITY:
Inclusion Criteria:

1. Parents of students in primary and secondary school.
2. Parents must had primary school education or above.

Exclusion Criteria:

1. Parents cannot speak or read Chinese.
2. Parents have severe mental or physical illness.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Parent-child conflict | 2 weeks
  The efficacy of parent-child conflict resolution will be assessed by the conflict subscale of the Conflict in Parent-Child Relationships. Scoring is based on a 5-point Likert scale with higher total scores indicate high level of conflict in the parent - child relationship.
Parent-child communication | 2 weeks
  The efficacy of communication, will be assessed by the family communication scale. Scoring is based on a 5-point Likert scale with regard to the quality of parent-child interactions. Higher total scores on individual and combined subscales indicate more positive parent-child interactions.
Parent-child Relationship | 2 weeks
  The efficacy of parent-child relationship intervention will be assessed by the parent-child relationship scale. Higher total scores indicate higher quality of parent-child relationship.
Couple Relationship Quality | 2 weeks
  The efficacy of Couple Relationship Intervention will be assessed by the quality of marriage index. Higher total scores indicate higher quality of couple relationship.
Marital Stability | 2 weeks
  The efficacy of Couple Relationship Intervention will be assessed by the stability of marriage scale-short form. Higher total scores indicate higher stability of couple relationship.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Normal University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No